CLINICAL TRIAL: NCT06932211
Title: A Study to Measure the Effect of a Toothpaste Containing Proteins and Enzymes and a Fluoride Toothpaste on Gingival Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ORL-GUM-3328
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Gingival Inflammation; Dental Plaque
MeSH Terms: conditions — Gingivitis; Dental Plaque | interventions — Enzymes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Statistician
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Test toothpaste (Experimental): Toothpaste containing proteins, enzymes and 1450 ppm fluoride as sodium fluoride
  Interventions: Other: Toothpaste containing proteins and enzymes
- Negative control toothpaste (Active Comparator): Toothpaste containing 1450 ppm fluoride as sodium fluoride
  Interventions: Other: Control fluoride toothpaste

INTERVENTIONS:
Other: Toothpaste containing proteins and enzymes — Toothpaste containing proteins, enzymes and 1450 ppm fluoride as sodium fluoride
  Arms: Test toothpaste
Other: Control fluoride toothpaste — Toothpaste containing sodium fluoride at 1450 ppm F
  Arms: Negative control toothpaste

SUMMARY:
This study is a double-blind, randomised, parallel group efficacy study. A minimum of 240 healthy female and male participants aged 18-70 years will be enrolled onto the study according to the inclusion/exclusion criteria. The accepted participants will then be randomly allocated to one of the two test products which they will use at home, twice a day for the duration of the study. Dental assessments of gingival condition and plaque level will be conducted after 4, 13 and 26 weeks of product use at the study site.

ELIGIBILITY:
Inclusion Criteria:

* Be in good general health.
* Be willing and physically able to carry out all study procedures.
* Be willing and competent (verbally and cognitively) to give written informed consent and complete a medical history form.
* Have at least 20 natural teeth without subgingival calculus including 5 teeth (excluding 3rd molars) in each quadrant, which can be assessed.
* Have mean Gingival Index (GI) score between 1.0 and 2.0 (1.0 ≤ Mean GI ≤ 2.0) and mean Plaque Index (PI) ≥ 1.5 at screening and baseline.
* Not have had a scale and prophylaxis in the month prior to enrolment or have one scheduled prior to the end of the study.
* Be willing to use only the test products for 6 months, after brushing with the products on site.
* Brush teeth twice daily (once in the morning and once at night).

Exclusion Criteria:

* Pregnant or breast feeding mothers.
* Subjects who participated in gum health study within 3 months prior to screening.
* Current participation in any other cosmetic trials, any dental clinical trials or clinical trials.
* Subjects who have used gum health products in the 4 weeks prior to screening.
* Obvious signs of untreated caries or significant periodontal disease, which in the opinion of the study dentist, will affect either the scientific validity of the study or if the participant was to participate in the study would affect their wellbeing.
* Full or partial dentures wearers.
* Current orthodontic treatment.
* Smokers or those who have a recent smoking history, including e-cigarettes.
* Diabetics.
* Medical condition and/or regular use of any medication which might affect the outcome of the study, as determined by the study dentist, principally a course of anti-inflammatory, antimicrobial or statin drugs within 4 weeks of screening.
* Taking dietary supplements (e.g. multivitamins, antioxidants, fish oils, etc.).
* Vegetarians and Vegans.
* Allergic to any ingredient of study products.
* The subject is a Unilever employee or a member of the study team.
* Any participant who, in the judgement of the investigator, should not participate in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 251 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2019-04-30 (Actual); Study Completion 2019-04-30 (Actual)

PRIMARY OUTCOMES:
Change in gingival condition as measured by Gingival Index | 13 weeks
  The gingival condition was assessed using gingival index (GI) [1]. The scoring criteria were: 0 = Absence of inflammation; 1 = Mild inflammation - slight change in colour and little change in texture; 2 = Moderate inflammation - moderate glazing, redness, oedema, and hypertrophy (bleeding on pressure); 3 = Severe inflammation - marked redness and hypertrophy (tendency to spontaneous bleeding). Each eligible tooth was scored at six sites: facial (body, mesial, distal) and lingual (body, mesial, distal). The participant's score at each timepoint is the average of all tooth sites measured.
  [1] LOE H, SILNESS J. Acta Odontol Scand. 1963;21:533-551.

SECONDARY OUTCOMES:
Change in gingival condition as measured by Gingival Index | 4 weeks and 26 weeks
  The gingival condition was assessed using gingival index (GI) [1]. The scoring criteria were: 0 = Absence of inflammation; 1 = Mild inflammation - slight change in colour and little change in texture; 2 = Moderate inflammation - moderate glazing, redness, oedema, and hypertrophy (bleeding on pressure); 3 = Severe inflammation - marked redness and hypertrophy (tendency to spontaneous bleeding). Each eligible tooth was scored at six sites: facial (body, mesial, distal) and lingual (body, mesial, distal). The participant's score at each timepoint is the average of all tooth sites measured.
  [1] LOE H, SILNESS J. Acta Odontol Scand. 1963;21:533-551.
Change in plaque levels as measured by Modified Quigley and Hein Plaque Index | 4 weeks, 13 weeks and 26 weeks
  Plaque was disclosed and assessed using modified Quigley and Hein plaque index (MQHPI) [1]. The scoring criteria were: 0 = No plaque; 1 = Separate flecks of plaque at the cervical margin of the tooth; 2 = A thin continuous band of plaque (up to one mm) at the cervical margin of the tooth; 3 = A band of plaque wider than one mm but covering less than 1/3 of the crown of the tooth; 4 = Plaque covering at least one-third but less than 2/3 of the crown of the tooth; 5 = Plaque covering 2/3 or more of the crown of the tooth. Each eligible tooth was scored at six sites: facial (body, mesial, distal) and lingual (body, mesial, distal). The participant's score at each timepoint is the average of all tooth sites measured.
  [1] Turesky S, Gilmore ND, Glickman I. J Periodontol. 1970;41(1):41-43.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Stomatology, Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No
Consent was not obtained from participants for this purpose.

REFERENCES:
- [Derived] Hu X, Zhang P, Zhang L, Matheson JR, Lin S, Sun JN, Delfanti C, Tian J, Gupta AK, Vasantharaghavan R, Huang R. The effect of enzyme and protein containing toothpaste on gingival condition: a randomised controlled study. BMC Oral Health. 2025 Nov 3;25(1):1727. doi: 10.1186/s12903-025-07096-7. PMID 41184910